CLINICAL TRIAL: NCT03137329
Title: Comparison of Surgical vs. Lifestyle Weight Treatment in Obese Older Adults
Brief Title: Surgical vs. Lifestyle in Obese Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not meet enrollment requirements with limited funding
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Christina Wee, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000188
Record Dates: First submitted 2017-03-27; First posted 2017-05-02 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Resistance Training; Nutritional Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight Loss Surgery (WLS) Arm (Other): Subjects enrolled in the WLS arm will undergo WLS as part of the routine care provided by the respective WLS centers. During routine care patients typically meet with their dietician at least twice prior to WLS and are placed on a higher protein meal replacement supplement and calorie controlled diet. For weeks 1-52, the investigators will ensure that patients are receiving 1500mg of elemental calcium and 3000 IU of vitamin D based on recent best practice guidelines. In addition, participants will complete an individualized pragmatic exercise program for the first 52 weeks after surgery. Patients will begin the program after receiving clearance from their surgeon. Patients will meet with a physical therapist at BIDMC for individual sessions.
  Interventions: Behavioral: Exercise program; Procedure: WLS
- Lifestyle Arm (Other): Subjects enrolled in the lifestyle group will be prescribed a balanced high protein diet (1g high quality protein/kg body weight/day) that provides an energy deficit of 500 to 750 kcal /day from their daily energy requirements[58] and prescribed a weight loss goal of 10% over the course of 6 months. Participants will meet with a trained dietician/nutritionist at the BIDMC General Clinical Research Unit. The investigators will incorporate the HMR (Health Management Resources) high protein meal replacement supplements into participants' diet regimen for the first 24 weeks. In addition, participants will complete a comparable 52-week exercise program consisting of an individualized pragmatic exercise program.
  Interventions: Behavioral: Exercise program; Dietary Supplement: Nutrition

INTERVENTIONS:
Behavioral: Exercise program — Physical therapy for aerobic and resistance training exercises
Dietary Supplement: Nutrition — Nutrition supplementation via HMR for lifestyle arm only
  Arms: Lifestyle Arm
Procedure: WLS — Weight loss surgery as planned
  Arms: Weight Loss Surgery (WLS) Arm

SUMMARY:
The study aims are

1. to demonstrate the feasibility of recruiting and enrolling 10 subjects aged 55-75 planning to undergo sleeve gastrectomy and enrolling 10-20 (1-2 per surgical patient) matched subjects to the described intensive lifestyle intervention.
2. to collect preliminary data on the comparative effectiveness of the two interventions on physical function, weight loss, body composition, bone density and QOL.

DETAILED DESCRIPTION:
The investigators propose a 1-year pilot feasibility study to examine the comparative effectiveness of sleeve gastrectomy compared to an intensive lifestyle intervention of a high protein low carbohydrate, hypocaloric weight loss diet combined with exercise training among older adults aged 60-75. For pragmatic and ethical reasons, the investigators are employing a nonrandomized design. The investigators will recruit 10 older patients undergoing sleeve gastrectomy and match, recruit, and enroll 1-2 subjects to the lifestyle intervention for each surgical subject. The investigators will assess physical function, weight loss, body composition, bone density, QOL and adverse events/health utilization at baseline and 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged 55-75 at the time of recruitment,
* speak English,
* meet medical eligibility criteria for WLS (i.e. BMI of >40 or >35 with a major obesity comorbidity),
* and be willing and able to participate in study procedures including the physical activity intervention and complete follow-up.

Exclusion Criteria:

The investigators will exclude participants for whom

* intentional weight loss might be inappropriate (e.g. patients with serious life-limiting illness)
* or who might be psychologically unstable (e.g. moderate to severe depression on the PHQ-9)
* or who have contraindications to a high protein diet or the physical activity intervention (e.g. recent MI/CVA in last 6 months, uncontrolled congestive heart failure, serum creatinine > 2.0 mg/dl/on dialysis, h/o celiac disease/crohn's disease/ulcerative colitis.)
* or patients whose weight exceeds 450 lbs (weight limit of DXA).
* The investigators will withdraw bariatric subjects who do not undergo weight loss surgery and his or her matched lifestyle subject. The investigators will withdraw subjects in the lifestyle group who do not attend at least attend two of the first three nutrition and physical therapy visits. The investigators will recruit additional subjects to replace lifestyle subjects who are withdrawn from the study for this reason.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Change in Physical Function | Years 1 and 2
  The primary outcome will be change in physical function as measured change in score on the Short Physical Performance Battery (SPPB) between the two groups at 6 months and 12 months. Secondary physical function outcomes includes change in performance on the Timed 400m walk and the sum of the one-repetition maximal weight subjects are able to lift in the biceps curl, bench press, seated row, knee extension and flexion, and leg press.[

SECONDARY OUTCOMES:
Change in anthropometric measurements-body weight | Years 1 and 2
  Changes in: body weight
Change in anthropometric measurements-waist circumference | Years 1 and 2
  Changes in: waist circumference
Change in body composition | Years 1 and 2
  Change in: fat mass, lean body mass of the whole body
Change in bone mineral density | Years 1 and 2
  Change in: bone density at the total hip and radius as measured by dual energy x-ray absorptiometry (DEXA) among subjects who weigh up to 450 lbs (equipment weight limit)
Change in blood pressure | Years 1 and 2
  Change in: blood pressure
Change in biochemical assessments-hbA1C | Years 1 and 2
  Change in: hemoglobin A1c,
Change in biochemical assessments-insulin and glucose | Years 1 and 2
  Change in: insulin and fasting glucose (insulin resistance)
Change in biochemical assessments-bone and muscle metabolism | Years 1 and 2
  Change in: biomarkers related to bone and muscle metabolism including vitamin D and bone alkaline phosphatase
Change in quality of life | Years 1 and 2
  Change in: Quality of life scores as measured by the Impact of Weight on Quality of Life and the Short Form-36
Change in pain | Years 1 and 2
  Change in: pain score using the Brief Pain Inventory
Change in disability | Years 1 and 2
  Change in: difficulty performing ADLs and IADLs
Change in medical history, medications and healthcare utilization from adverse events | Years 1 and 2
  all visits, hospitalizations, and emergency room visits including any study related visits.

CONTACTS AND LOCATIONS:
Overall Officials: Christina C Wee, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No